CLINICAL TRIAL: NCT04644666
Title: Incidence and Risk Factors for Persistent Post-sternotomy Pain After Cardiac Surgery in Local Chinese Population: a Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, WONG MAN KIN, Honorary Clinical Associate Professor, Associate Consultant, Chinese University of Hong Kong
Other Study IDs: 2020.446-T
Record Dates: First submitted 2020-11-17; First posted 2020-11-25 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CPSP is common after cardiac surgery. The reported incidence was 28% to 56% up to 2 years postoperatively. Despite a large number of cross-sectional and retrospective studies, prospective cohort studies examining the incidence of chronic post-sternotomy pain following cardiac surgery have been scarce, and none on our local Chinese population.

Several mechanisms have been involved in the development of chronic pain after sternotomy. Ongoing pain after surgery can continue to sensitize the nociceptive fibres which may subsequently lead to hyperalgesia, hyperpathia, allodynia and dysesthesia. In addition, like any form of chronic pain, it is a multidimensional process involving social, cognitive and psychological factors.

CPSP has the potential to impact daily functioning and quality of life of patients, as well as increasing the healthcare costs. To date, only the CARDpain study examined the role of social and psychological risk factors in development of CPSP after cardiac surgery. They found pre-surgical anxiety, measured by the Hospital and Anxiety Depression Scale (HADS), was a significant risk factor.

The primary aim of the study is to examine the incidence of chronic post-sternotomy pain at 3 months and 6 months following cardiac surgery in local Chinese population, and identify the clinical and psychological risk factors associated with its development. The secondary aim is to determine the impact of CPSP on the quality of life following cardiac surgery.

DETAILED DESCRIPTION:
Postoperative pain that persists beyond the normal time for tissue healing is increasingly recognized as an important complication after various types of surgery. According to the International Association for Study of Pain (IASP), chronic postsurgical pain (CPSP) is defined as the persistence of pain at surgical site or referred area, at least 3 months following the surgical procedure1. CPSP is common after cardiac surgery. The reported incidence was 28% to 56% up to 2 years postoperatively. The wide range of reported incidence seems to result from heterogenicity of the study population and the study design. McGillion MH et al reviewed that cross-sectional and retrospective studies have generally reported higher prevalence for CPSP (14-56%) after cardiac surgery than those investigations with prospective designs (7.5-45%). Despite a large number of cross-sectional and retrospective studies, prospective cohort studies examining the incidence of chronic post-sternotomy pain following cardiac surgery have been scarce, and none on our local Chinese population.

Several mechanisms have been involved in the development of chronic pain after sternotomy. These include dissection, nerve entrapment by sternal wires, sternal retraction which can dislocate and fractured ribs, and intercostal neuralgia as a consequence of nerve damage during dissection of the internal mammary artery during coronary artery bypass graft (CABG). All can stimulate the release of proinflammatory cytokines which sensitize the afferent nociceptive fibres to cause chronic pain. Ongoing pain after surgery can continue to sensitize the nociceptive fibres which may subsequently lead to hyperalgesia, hyperpathia, allodynia and dysesthesia. In addition, like any form of chronic pain, it is a multidimensional process involving social, cognitive and psychological factors.

CPSP has the potential to impact daily functioning and quality of life of patients, as well as increasing the healthcare costs. CARDpain study reported that among those with CPSP, over 50% had significant pain-related interference with activities of daily living (family and home responsibilities, recreation and employment) at 3, 6 and 12 months following cardiac surgery. Identification of risk factors associated with the development of CPSP could potentially improve outcomes among high-risk patients, especially if the risk factors are modifiable. To date, only the CARDpain study examined the role of social and psychological risk factors in development of CPSP after cardiac surgery. They found pre-surgical anxiety, measured by the Hospital and Anxiety Depression Scale (HADS), was a significant risk factor.

The primary aim of our study is to examine the incidence of chronic post-sternotomy pain at 3 months and 6 months following cardiac surgery in our local Chinese population, and identify the clinical and psychological risk factors associated with its development. The secondary aim is to determine the impact of CPSP on the quality of life following cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 or older
2. Elective surgery
3. Primary isolated coronary artery bypass grafting, aortic valve repair/replacement or combined coronary artery bypass/valve procedure via sternotomy for the first time

Exclusion Criteria:

1. Emergency surgery
2. Redo surgery
3. History of thoracotomy or mastectomy
4. History of psychosis or illicit drug use
5. Estimated glomerular filtration rate (eGFR) <30ml/min or on renal replacement therapy. This is calculated using Cockcroft-Gault formula
6. Intraoperative use of remifentanil
7. Unable to provide informed consent and complete the questionnaires because of physical or mental incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Local Chinese population age 18 or older undergoing elective open heart surgery
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic post-sternotomy pain in number | 3 months after surgery
  Number of recruited patients who have chronic pain
Incidence of chronic post-sternotomy pain in percentage | 3 months after surgery
  Percentage of recruited patients who have chronic pain
Incidence of chronic post-sternotomy pain | 6 months after surgery
  Number of recruited patients who have chronic pain
Incidence of chronic post-sternotomy pain | 6 months after surgery
  Percentage of recruited patients who have chronic pain

SECONDARY OUTCOMES:
Association between the severity of acute postoperative pain (measured using visual analogue scale) and the presence of chronic post-surgical pain | Acute postoperative pain captured within 72 hours and on Day 7 after surgery using visual analogue score
  Pain score assessment using visual analogue scale. The score ranges from 0 to 10. The severity of pain increases with the score. Statistical analysis will be used to identify the associate between acute pain and chronic post-surgical pain in cardiac surgical patients.
Association between the amount of intraoperative and postoperative opioid consumption and the presence of chronic post-surgical pain | Opioid consumption during surgery and within 72 hours after surgery will be captured
  Total opioid consumption intraoperatively and postoperatively in ICU and ward will be recorded. Intraoperative opioid consumption can be extracted from the anesthetic record. Postoperative opioid consumption can be recorded from the Patient-controlled Analgesia machine. The dose of all opioids used will be converted into morphine equivalent dose. Regression analysis will be used to identify the relationship between opioid consumption and chronic post-surgical pain in cardiac surgery
Association between psychological risk factors and chronic post-surgical pain | Hospital Anxiety and Depression Scale will be assessed 1 day before surgery, 3 month postop and 6 month postop
  Psychological risk factors assessed using Hospital Anxiety and Depression Scale
Association between psychological risk factors and chronic post-surgical pain | EQ-5D questionnaire will be assessed 1 day before surgery, 3 month postop and 6 month postop
  Quality of life will be assessed using EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong